CLINICAL TRIAL: NCT05871411
Title: Validation of Visual Analog Scales to Measure SatisfactiOn and WELL-being at Work (SoWell-VAS)
Acronym: SoWell-VAS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2022 DUTHEIL; 2022-A02450-43 (Other: 2022-A02450-43)
Record Dates: First submitted 2023-05-03; First posted 2023-05-23 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Validation; Visual Analogue Scale; Occupational Stress
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We spend a third of our life at work. Psychosocial risks (PSR) are a major issue in occupational health 1. Approaching the different dimensions of PSR calls on a dozen essential components: workload, autonomy, social support, burnout, anxiety, efforts made, rewards, work addiction, investment, etc. a specific questionnaire which usually contains 20 to 30 questions, so that having an overall view of PSR using the current reference questionnaires (Karasek, Siegrist, etc.) represents a total of more than 300 questions. The response time is thus incompatible with current medical practice (passage in the waiting room before the occupational health medical examination) and leads to a majority of non-responses during anonymous questionnaires on the Internet. On the other hand, these validated questionnaires were carried out by different people and are very heterogeneous between them, including in their formulation, so that the respondents have the impression of disorganization and anarchy. There is therefore a need for short, quick and uniform questionnaires. EVAs offer the incredible advantage of meeting these criteria: speed, uniformity, precision. From a data analysis point of view, EVAs also have the advantage of offering a continuous quantitative response, allowing the use of all statistical approaches. If some questionnaires have already been validated in the form of EVA, such as the EVA stress versus the " Perceived Stress Scale " questionnaire (PSS), the EVA workload and EVA autonomy at work versus the Karasek questionnaire, the other reference questionnaires are not yet validated in EVA (burnout, anxiety, efforts / rewards, work addiction, etc.).

ELIGIBILITY:
Inclusion Criteria:

* All voluntary adults with a professional activity.

Exclusion Criteria:

* Minor
* Person not volunteer to participate.
* Protected adults (curatorship, guardianship, safeguard of justice)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with a professional activity
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Burnout | Inclusion
  Burnout on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Burnout | One week later
  Burnout on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Burnout | Inclusion
  Burnout using the Maslach Burn-out Inventory (MBI) questionnaire. MBI is composed of 22 items designed to assess the three components of the burn-out syndrome: emotional exhaustion (9 items), depersonalization (5 items) and reduced personal accomplishment (8 items). The items are written in the form of statements about personal feelings or attitudes. Items are made of a 7-point scale frequency of feelings, varying from "never" to "every day". The scores for each component of the burn-out syndrome are considered separately and are not combined into a single total score. If desired for participant feedback, each score can be coded as low, average, or high
Burnout | One week later
  Burnout using the Maslach Burn-out Inventory (MBI) questionnaire. MBI is composed of 22 items designed to assess the three components of the burn-out syndrome: emotional exhaustion (9 items), depersonalization (5 items) and reduced personal accomplishment (8 items). The items are written in the form of statements about personal feelings or attitudes. Items are made of a 7-point scale frequency of feelings, varying from "never" to "every day". The scores for each component of the burn-out syndrome are considered separately and are not combined into a single total score. If desired for participant feedback, each score can be coded as low, average, or high
Anxiety | Inclusion
  Anxiety on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Anxiety | One week later
  Anxiety on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Anxiety | Inclusion
  Anxiety using Hospital Anxiety and Depression (HAD) questionnaire. is a self-reported questionnaire composed of 14 items with a 4-point Likert scale assessing anxiety (7 items) and/or depressive (7 items) symptoms. For each subscale (anxiety and depression), total score ranges from 0 to 21. Higher scores indicate higher levels of anxiety or depressive symptoms. A score from 0 to 7 indicates the absence of disease, a score of 8-10 represents doubtful cases, and scores higher than 11 reflects the presence of a mood disorder.
Anxiety | One week later
  Anxiety using Hospital Anxiety and Depression (HAD) questionnaire. is a self-reported questionnaire composed of 14 items with a 4-point Likert scale assessing anxiety (7 items) and/or depressive (7 items) symptoms. For each subscale (anxiety and depression), total score ranges from 0 to 21. Higher scores indicate higher levels of anxiety or depressive symptoms. A score from 0 to 7 indicates the absence of disease, a score of 8-10 represents doubtful cases, and scores higher than 11 reflects the presence of a mood disorder.
Job demand | Inclusion
  Job demand on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Job demand | One week later
  Job demand on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Job control | Inclusion
  Job control on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Job control | One week later
  Job control on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Social support | Inclusion
  Social support on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Social support | One week later
  Social support on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Job demand / job control / social support | Inclusion
  Job demand / job control / social support using the Job Demand-Control-Support (JDSC) questionnaire of Karasek. JDSC assessed job demands, job control and social support through 26 items. The questionnaire measures nine items of job demands, nine items of job control and eight items of social support. Items of JDSC are scored on a four-point Likert-type scale, ranging from 1 = strongly disagree to 4 = strongly agree. Among the 26 items, five negative statements require reverse scoring. From French data, the job strain threshold is set for a demands score higher than 20 and a control score lower than 71; the isostrain threshold is determined from a combining score of job strain and social support lower than 24.
Job demand / job control / social support | One week later
  Job demand / job control / social support using the Job Demand-Control-Support (JDSC) questionnaire of Karasek. JDSC assessed job demands, job control and social support through 26 items. The questionnaire measures nine items of job demands, nine items of job control and eight items of social support. Items of JDSC are scored on a four-point Likert-type scale, ranging from 1 = strongly disagree to 4 = strongly agree. Among the 26 items, five negative statements require reverse scoring. From French data, the job strain threshold is set for a demands score higher than 20 and a control score lower than 71; the isostrain threshold is determined from a combining score of job strain and social support lower than 24.questionnaire of Karasek
Effort-reward imbalance | Inclusion
  Effort-reward imbalance on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Effort-reward imbalance | One week later
  Effort-reward imbalance on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Effort-reward imbalance | Inclusion
  Effort-reward imbalance using Effort-Reward Imbalance Questionnaire (ERI). ERI assessed psychological distress and health problems that may occur when there is an imbalance between the efforts required by the work and the rewards received. We used the 46 items of the French version of the ERI model exploring efforts (six items), over commitment (eleven items), and rewards (seventeen items). Items of ERI were scored on a five-point Likert-type scale, ranging from 1 = disagree to 5 = agree and very disturbed. A ratio extrinsic efforts and rewards can assess the imbalance between these two dimensions. A ratio greater than one defines employees exposed to an imbalance between efforts and rewards
Effort-reward imbalance | One week later
  Effort-reward imbalance using Effort-Reward Imbalance Questionnaire (ERI). ERI assessed psychological distress and health problems that may occur when there is an imbalance between the efforts required by the work and the rewards received. We used the 46 items of the French version of the ERI model exploring efforts (six items), over commitment (eleven items), and rewards (seventeen items). Items of ERI were scored on a five-point Likert-type scale, ranging from 1 = disagree to 5 = agree and very disturbed. A ratio extrinsic efforts and rewards can assess the imbalance between these two dimensions. A ratio greater than one defines employees exposed to an imbalance between efforts and rewards
Work addiction | Inclusion
  Work addiction on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Work addiction | One week later
  Work addiction on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Work addiction | Inclusion
  Work addiction using Work Addiction Risk Test (WART) questionnaire. The WART assesses 25 statements on a 4-point Likert scale from 1 - never true to 4 - always true. The total score ranged from 25 to 100, with higher scores reflecting higher work addiction. Scores from 25 to 56 were defined as low-risk of work addiction; from 57 to 66 as medium-risk and from 67 to 100 as high-risk .
Work addiction | One week later
  Work addiction using Work Addiction Risk Test (WART) questionnaire. The WART assesses 25 statements on a 4-point Likert scale from 1 - never true to 4 - always true. The total score ranged from 25 to 100, with higher scores reflecting higher work addiction. Scores from 25 to 56 were defined as low-risk of work addiction; from 57 to 66 as medium-risk and from 67 to 100 as high-risk .
Life satisfaction | Inclusion
  Life satisfaction on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Life satisfaction | One week later
  Life satisfaction on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Life satisfaction | Inclusion
  Life satisfaction using the Minnesota Satisfaction Questionnaire (MSQ). MSQ is composed of 20 items designed to measure employee job satisfaction. Items are made of a 5-point scale of satisfaction, varying from 1 "Very dissatisfied" to 5 "Very satisfied". A percentile score of 75 or higher represent a high degree of satisfaction, a percentile score of 25 or lower represent a low degree of satisfaction and scores in the middle range of percentiles (26 to 74) indicated average satisfaction.
Life satisfaction | One week later
  Life satisfaction using the Minnesota Satisfaction Questionnaire (MSQ). MSQ is composed of 20 items designed to measure employee job satisfaction. Items are made of a 5-point scale of satisfaction, varying from 1 "Very dissatisfied" to 5 "Very satisfied". A percentile score of 75 or higher represent a high degree of satisfaction, a percentile score of 25 or lower represent a low degree of satisfaction and scores in the middle range of percentiles (26 to 74) indicated average satisfaction.

SECONDARY OUTCOMES:
Sociodemographic | Once at inclusion
  age, gender, marital status, number of children, education level
Occupation | Once at inclusion
  Question "What is your profession?"
Work hours per week | Once at inclusion
  Number of hours worked per week
Night and weekend work | Once at inclusion
  Do you work at night? Do you work weekends?
Alcohol consumption | Once at inclusion
  Number of alcoholic drinks per week
Tabacco consumption | Once at inclusion
  Number of cigarettes per day
Height | Once at inclusion
  Height in cm
Weight | Once at inclusion
  Weight in kg
Sedentary behavior | Once at inclusion
  Number of hours sit per day
Physical activity | Once at inclusion
  Number of hours of physical activity per day
Stress at work | Once at inclusion
  stress at work level on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Ethical conflicts | Once at inclusion
  Ethical conflicts confrontation on a horizontal, non-calibrated line of 100 mm, ranging from never (0) to often(100)
Perceived health | Once at inclusion
  Perceived health on a horizontal, non-calibrated line of 100 mm, ranging from bad(0) to excellent (100)
Stress at home | Once at inclusion
  stress at home level on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Fatigue | Once at inclusion
  Fatigue level on a horizontal, non-calibrated line of 100 mm, ranging from minimum (0) to maximum (100)
Sleep quality | Once at inclusion
  Sleep quality level on a horizontal, non-calibrated line of 100 mm, ranging from bad(0) to excellent (100)
Mood | Once at inclusion
  mood level on a horizontal, non-calibrated line of 100 mm, ranging from bad(0) to excellent (100)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Dutheil, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Clinchamps M, Pereira B, Mermillod M, Charkhabi M, Zak M, Jiao J, Cole A, Bouillon-Minois JB, Dutheil F. Validation of visual analogue scales to assess occupational stress compared to the Karasek questionnaire: A cross sectional study. PLoS One. 2026 Feb 10;21(2):e0340209. doi: 10.1371/journal.pone.0340209. eCollection 2026. PMID 41666222